CLINICAL TRIAL: NCT04232878
Title: A Phase 1, Double-Blind, Sponsor-Open, Placebo-Controlled, First-In-Human Trial To Evaluate The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Single Ascending Doses of CVL-936 In Healthy Subjects
Brief Title: A Single Ascending Dose Trial of CVL-936 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sufficient data has been obtained to meet current objectives
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVL-936-HV-001
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Substance Use Disorders (SUD)
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: A sample size of 9 subjects per cohort has been chosen based on the need to minimize exposure of humans to CVL-936 and PF-06815106 and the requirement to provide adequate safety, tolerability, and PK information at each dose. Each cohort will be conducted as a crossover design with 3 periods and each cohort will have up to 6 subjects receiving CVL-936 and 3 subjects receiving placebo within each period, with a total of approximately 18 subjects if 2 cohorts complete or a total of approximately 27 subjects if 3 cohorts complete.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Active Comparator: Group 1 Period 1: 0.5mg CVL-936 (Active Comparator): Oral suspension/solution
  Interventions: Drug: CVL-936
- Placebo Comparator: Group 1 Period 1: 0.5mg Matching Placebo (Placebo Comparator): Matching Placebo; Oral suspension/solution
  Interventions: Drug: Matching Placebo
- Active Comparator: Group 1 Period 2:TBD mg CVL-936 (Active Comparator): Oral suspension/solution
  Interventions: Drug: CVL-936
- Placebo Comparator: Group 1 Period 2:TBD mg Matching Placebo (Placebo Comparator): Matching Placebo; Oral suspension/solution
  Interventions: Drug: Matching Placebo
- Active Comparator: Group 1 Period 3:TBD mg CVL-936 (Active Comparator): Oral suspension/solution
  Interventions: Drug: CVL-936
- Placebo Comparator: Group 1 Period 3:TBD mg Matching Placebo (Placebo Comparator): Matching Placebo; Oral suspension/solution
  Interventions: Drug: Matching Placebo
- Active Comparator: Group 2 Period 1:TBD mg CVL-936 (Active Comparator): Oral suspension/solution
  Interventions: Drug: CVL-936
- Placebo Comparator: Group 2 Period 1:TBD mg Matching Placebo (Placebo Comparator): Matching Placebo; Oral suspension/solution
  Interventions: Drug: Matching Placebo
- Active Comparator: Group 2 Period 2:TBD mg CVL-936 (Active Comparator): Oral suspension/solution
  Interventions: Drug: CVL-936
- Placebo Comparator: Group 2 Period 2:TBD mg Matching Placebo (Placebo Comparator): Matching Placebo; Oral suspension/solution
  Interventions: Drug: Matching Placebo
- Active Comparator: Group 2 Period 3:TBD mg CVL-936 (Active Comparator): Oral suspension/solution
  Interventions: Drug: CVL-936
- Placebo Comparator: Group 2 Period 3:TBD mg Matching Placebo (Placebo Comparator): Matching Placebo; Oral suspension/solution
  Interventions: Drug: Matching Placebo
- Active Comparator: Group 3: TBD mg CVL-936 (Active Comparator): Oral suspension/solution
  Interventions: Drug: CVL-936
- Placebo Comparator: Group 3: TBD mg Matching Placebo (Placebo Comparator): Matching Placebo; Oral suspension/solution
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: CVL-936 — CVL-936
  Arms: Active Comparator: Group 1 Period 1: 0.5mg CVL-936; Active Comparator: Group 1 Period 2:TBD mg CVL-936; Active Comparator: Group 1 Period 3:TBD mg CVL-936; Active Comparator: Group 2 Period 1:TBD mg CVL-936; Active Comparator: Group 2 Period 2:TBD mg CVL-936; Active Comparator: Group 2 Period 3:TBD mg CVL-936; Active Comparator: Group 3: TBD mg CVL-936
Drug: Matching Placebo — Placebo matching CVL-936
  Arms: Placebo Comparator: Group 1 Period 1: 0.5mg Matching Placebo; Placebo Comparator: Group 1 Period 2:TBD mg Matching Placebo; Placebo Comparator: Group 1 Period 3:TBD mg Matching Placebo; Placebo Comparator: Group 2 Period 1:TBD mg Matching Placebo; Placebo Comparator: Group 2 Period 2:TBD mg Matching Placebo; Placebo Comparator: Group 2 Period 3:TBD mg Matching Placebo; Placebo Comparator: Group 3: TBD mg Matching Placebo

SUMMARY:
The aim of this trial is to investigate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of CVL-936 following single ascending oral doses in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects and female subjects of nonchildbearing potential, ages 18 to 50 years

Exclusion Criteria:

1. Subjects with a current history of significant pulmonary, gastrointestinal, renal, hepatic, metabolic, endocrine, hematological, immunological, psychiatric, or neurological disease that, in the opinion of the investigator or medical monitor, could compromise either subject safety or the results of the trial.
2. Subjects with epilepsy or a history of seizures
3. Systolic supine blood pressure ≥130 mmHg and/or supine diastolic blood pressure ≥80 mmHg at Screening or Day -1, or orthostatic hypotension at Screening or Day -1.
4. Subjects with a history of hypersensitivity to any dopamine-blocker medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with reported Treatment Emergent Adverse Events (TEAEs) | At the end of Period 3 (30 Days)
Number of Subjects with Clinically significant changes in Electrocardiogram measures (PR, RR, QT and QTcF) | At the end of Period 3 (30 Days)
Number of Subjects with Clinically meaningful changes in Vital signs (Systolic and Diastolic blood pressures, heart rate, respiratory rate and body temperature) | At the end of Period 3 (30 Days)
Number of Subjects with Clinically significant changes in laboratory measures | At the end of Period 3 (30 Days)
  Number of subjects with clinically significant changes in hematology, serum chemistry and urinalysis will be reported
Change from baseline of the Columbia-Suicide Severity Rating Scale (C-SSRS) | At the end of Period 3 (30 Days)
  The C-SSRS rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent).
Change from Baseline of Simpson-Angus Scale (SAS) Results | At the end of Period 3 (30 Days)
  Evaluating Extrapyramidal symptoms using the SAS. The SAS consists of a list of 10 symptoms of parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia). Each item is rated on a 5-point scale, with a score of 0 representing absence of symptoms and a score of 4 representing a severe condition. The SAS total score is the sum of the scores for all 10 items.
Change from Baseline of Abnormal Involuntary Movement Scale (AIMS) Results | At the end of Period 3 (30 Days)
  The AIMS assessment consists of 10 items describing symptoms of dyskinesia. Facial and oral movements (items 1 through 4), extremity movements (items 5 and 6), and trunk movements (item 7) are observed unobtrusively while the subject is at rest, and the investigator also makes global judgments on the subject's dyskinesias (items 8 through 10). Each item is rated on a 5-point scale, with a score of 0 representing absence of symptoms (for item 10, no awareness), and a score of 4 indicating a severe condition (for item 10, awareness, severe distress). In addition, the AIMS includes 2 yes/no questions that address the subject's dental status. The AIMS Movement Rating Score is defined as the sum of items 1 through 7 (ie, items 1 through 4, facial and oral movements; items 5 and 6, extremity movements; and item 7, trunk movements).
Change from Baseline of Barnes Akathisia Rating Scale (BARS) Results | At the end of Period 3 (30 Days)
  Evaluating Extrapyramidal symptoms using the BARS. The BARS consists of 4 items related to akathisia: objective observation of akathisia by the investigator, subjective feelings of restlessness by the subject, subjective distress due to akathisia, and global clinical assessment of akathisia. The first 3 items are rated on a 4-point scale, with a score of 0 representing absence of symptoms and a score of 3 representing a severe condition. The global clinical evaluation is made on a 6-point scale, with a score of 0 representing absence of symptom and a score of 5 representing severe akathisia.

CONTACTS AND LOCATIONS:
Overall Officials: Matt Leoni, MD, Study Director — Cerevel Therapeutics, LLC
Locations (1):
- Hassman Research Institute, Marlton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No